CLINICAL TRIAL: NCT01721278
Title: A Prospective Multicentre Clinical Surveillance Study To Evaluate The Stability, Efficacy And Safety Of The Furlong Evolution® Hip Stem In Primary Total Hip Arthroplasty
Brief Title: Furlong Evolution® Hip Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Joint Replacement Instrumented Orthopaedics Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: 12/LO/0768
Record Dates: First submitted 2012-10-16; First posted 2012-11-05 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Focus: A Multicentre Prospective Clinical Surveillance Study Aims to Assess the Clinical, Functional and Radiological Outcome of the Furlong Evolution® Hip Stem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Total hip replacement (THR) is a highly effective procedure in relieving pain and restoring function. Many different implants can be used in artificial hip joints. Hydroxyapatiteceramic (HAC) coating has become a well established The JRI Furlong® HAC femoral stem is one such implant with good long term survivorship. The femoral implant has been used since 1985 and published findings have shown a 97.4% survivorship at a mean of 17 years follow up in patients. The Furlong Evolution® design is based on the tried and tested Furlong HAC but with some modifications.

This is a 10 year multicentre clinical surveillance study, which aims to assess the clinical, functional and radiological performance of the Furlong Evolution® Hip stem in human patients.

DETAILED DESCRIPTION:
Purpose and Design:

The Furlong Evolution® design is based on the tried and tested Furlong H.A.C implant but with some modifications. It still retains its full H.A.C coating and is much shorter in length. This potentially makes it easier to introduce into the femoral canal, which may result in less soft tissue damage and lower rate of femoral fracture. This would be very beneficial, should revision (implant replacement) be required at a later date. This potential characteristic has been highlighted as an important component of determining the clinical effectiveness of a total hip replacement.

As per the National Institute of Clinical Excellence (NICE) guidelines the best prostheses demonstrates a revision rate (the rate at which they need to be replaced) of 10% or less at 10 years. This should be regarded as the current benchmark in the selection of prostheses for primary Total Hip Replacement (THR). It is also considered reasonable to recommend a prostheses with a maximum of 3% revision rate at 3 years which would indicate performance would then be subjected to annual review (up to 10 years) to ensure that the revision rate remains consistent with the 10year benchmark. The Orthopaedic Data Evaluation Panel (ODEP) was established to evaluate data on the outcomes of prostheses provided by manufactures and to inform the NHS which products are compliant with the benchmarks set by NICE. Therefore this study will be a ODEP compliant multicentre prospective surveillance study of the Furlong Evolution® Hip Stem that will assess the clinical, functional and radiographical performance over a 10 year period in compliance with the NICE guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. All patients consenting to total hip replacement
2. All patients deemed suitable for total hip replacement
3. All patients passing pre-assessment deeming them medically fit enough for total hip replacement.

Exclusion Criteria:

1. Patients deemed unsuitable for Total Hip Replacement
2. Patients who refuse to have surgery opting for other modes of treatment
3. Patients who are unable to consent due to a lack of capacity
4. Patients unable to understand English
5. Any patient under the age of 18 years.
6. Patients who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As per ODEP guidelines, a minimum of 500 cohort size is required for benchmark validation of the clinical performance of a new orthopaedic implant. We will be using a total sample size of 700 patients over 10 centres to ensure we meet the benchmark validation criteria.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2012-10; Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
The performance of the Furlong Evolution Hip Stem will be assessed clinically and radiographically of all participants. Number of participants who have reported complications, adverse events & serious adverse events will act as a measure of safety. | 10 years

SECONDARY OUTCOMES:
Questionnaires (Oxford Hip,EQ5D & Harris Hip Score) will be obtained from participating subjects to evaluate patient function & satisfaction & quality of life at each follow up visit. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Professor Justin Cobb, MCh FRCS, Principal Investigator — Imperial College London
Locations (1):
- Charing Cross hospital, London, United Kingdom